CLINICAL TRIAL: NCT01038778
Title: Phase I/II Study of High Dose Interleukin 2, Aldesleukin, in Combination With the Histone Deacetylase Inhibitor Entinostat in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Entinostat in Combination With Aldesleukin in Treating Patients With Metastatic Kidney Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02900; NCI-2012-02900 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000662915; I 145208; 7870 (Other: Roswell Park Cancer Institute); 7870 (Other: CTEP); P30CA016056 (NIH); R21CA137649 (NIH); U01CA062505 (NIH); U01CA070095 (NIH); U01CA076576 (NIH); UM1CA186691 (NIH); UM1CA186712 (NIH); UM1CA186717 (NIH); NCT01043159 (obsolete NCT alias)
Record Dates: First submitted 2009-12-18; First posted 2009-12-24 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Clear Cell Renal Cell Carcinoma; Metastatic Kidney Carcinoma; Stage III Renal Cell Cancer AJCC v7; Stage IV Renal Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — aldesleukin; entinostat; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (entinostat, aldesleukin) (Experimental): Patients receive entinostat PO every 2 weeks beginning on day -14 and high-dose aldesleukin IV every 8 hours on days 1-5 and 15-19. Cycles repeat every 84 days* in the absence of disease progression or unacceptable toxicity.
  NOTE: *Patients with evidence of tumor shrinkage may receive up to 3 cycles of high-dose aldesleukin therapy. Patients with stable disease by RECIST version 1.0 criteria, but without evidence of tumor shrinkage after two cycles will receive only entinostat until disease progression is documented.
  Interventions: Biological: Aldesleukin; Procedure: Computed Tomography; Drug: Entinostat; Radiation: Fludeoxyglucose F-18; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Aldesleukin — Given IV
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Procedure: Computed Tomography — Undergo FDG-PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; MS 27-275; MS 275; MS-275; MS275; SNDX 275; SNDX-275; SNDX275
Radiation: Fludeoxyglucose F-18 — Undergo FDG-PET/CT
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Procedure: Positron Emission Tomography — Undergo FDG-PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase I/II trial studies the side effects and best dose of entinostat when given together with aldesleukin and to see how well this works in treating patients with kidney cancer that has spread to other places in the body. Entinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Aldesleukin may stimulate the white blood cells to kill kidney cancer cells. Giving entinostat together with aldesleukin may be a better treatment for metastatic kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of high dose interleukin 2 (aldesleukin) in combination with entinostat in patients with metastatic renal cell carcinoma (RCC). (Phase I) II. To monitor toxicity and estimate the efficacy of high dose aldesleukin combined with entinostat in patients with metastatic RCC. (Phase II)

SECONDARY OBJECTIVES:

I. To compare the time-to-tumor progression, progression-free survival and overall survival of patients with metastatic RCC treated with high dose aldesleukin combined with entinostat to the historical data of patients treated with high dose aldesleukin alone. (Phase II) II. To assess the toxicity of high dose aldesleukin combined with entinostat. (Phase II) III. To evaluate entinostat pharmacodynamics (PD) in blood and tumor samples. (Phase II) IV. To measure the association between baseline laboratory parameters (e.g. cluster of differentiation [CD]4+, CD8+, CD4+/forkhead box P3 [Foxp3]), tumor blood metabolism, and a variety of response variables (e.g. toxicity, response and survival). (Phase II) V. To explore the relationship between entinostat exposure with PD endpoints (e.g. toxicity and histone acetylation in peripheral blood mononuclear cells or peripheral blood mononuclear cells [PBMNCs] and changes in T cell subset population). (Phase II) VI. To evaluate the modulation of tumor metabolism by fluorodeoxyglucose (FDG, fludeoxyglucose F 18) positron emission tomography (PET)/computed tomography (CT) scan. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of entinostat followed by a phase II study.

Patients receive entinostat orally (PO) every 2 weeks beginning on day -14 and high-dose aldesleukin intravenously (IV) every 8 hours on days 1-5 and 15-19. Cycles repeat every 84 days* in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients with evidence of tumor shrinkage may receive up to 3 cycles of high-dose aldesleukin therapy. Patients with stable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0 criteria, but without evidence of tumor shrinkage after two cycles will receive only entinostat until disease progression is documented.

After completion of study treatment, patients are followed up at 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathological diagnosis of renal cell carcinoma that is metastatic or surgically unresectable; the histology must be clear cell carcinoma or predominant clear cell carcinoma
* Patients may have received up to two prior therapies including vascular endothelial growth factor (VEGF), mammalian target of rapamycin (mTOR) and programmed cell death (PD)-1/PD ligand 1 (L1) inhibitors; prior palliative radiation to metastatic lesion(s) is permitted, provided there is at least one measurable and/or evaluable lesion(s) that has not been irradiated
* Patients must have measurable or evaluable disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0
* Life expectancy of greater than 6 months
* Hemoglobin >= 12 g/dL
* Leukocytes >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Total bilirubin =< 1.5 x laboratory upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x laboratory upper limit of normal
* Creatinine =< 1.5 x laboratory upper limit of normal or calculated creatinine clearance of >= 50 ml/min
* Lactate dehydrogenase (LDH) within normal limits (WNL)
* Corrected calcium =< 10 mg/dL
* Prothrombin time (PT)/international normalized ratio (INR) =< 1.5
* Urine protein < 1+; if >= 1+, 24 hour urine protein should be obtained and should be < 1000 mg
* Forced expiratory volume in 1 second (FEV1) >= 2.0 liters or >= 75% of predicted for height and age; (pulmonary function tests [PFTs] are required for patients over 50 or with significant pulmonary or smoking history)
* No evidence of congestive heart failure, symptoms of coronary artery disease, myocardial infarction less than 6 months prior to entry, serious cardiac arrhythmias, or unstable angina; patients who are over 40 or have had previous myocardial infarction greater than 6 months prior to entry will be required to have a negative or low probability cardiac stress test for cardiac ischemia
* No history of cerebrovascular accident or transient ischemic attacks
* The effects of entinostat on the developing human fetus at the recommended therapeutic dose are unknown; for this reason Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; men with female partners of child bearing potential must also agree to use adequate contraception
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have received more than two prior therapies
* Concurrent use of valproic acid is not allowed
* Patients may not be receiving any other investigational agents
* Patients with untreated central nervous system (CNS) metastases; patients should have a head CT/magnetic resonance imaging (MRI) within 28 days prior to treatment initiation; patients with previously excised/gamma knifed solitary or oligometastases and controlled disease are eligible
* Any medical condition that would preclude adequate evaluation of the safety and toxicity of the study combination
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Association class II, III, or IV), angina pectoris requiring nitrate therapy, recent myocardial infarction (< the last 6 months), cardiac arrhythmia, history of cerebrovascular accident (CVA) within 6 months, hypertension (defined as blood pressure of > 160 mmHg systolic and/or > 90 mmHg diastolic on medication) history of peripheral vascular disease, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with a history of allergy to entinostat or other medications that have a benzamide structure (i.e. tiapride, remoxipride, and clebopride)
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with entinostat
* Human immunodeficiency virus (HIV)-positive patients receiving combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with entinostat. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Serious or non-healing wound, ulcer or bone fracture
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 1 therapy
* Anticipation of need for major surgical procedures during the course of the study
* Left ventricular ejection function < 45%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-10-29 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2026-02-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Saby George, Principal Investigator — Roswell Park Cancer Institute
Locations (4):
- United States (4):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Roswell Park Cancer Institute, Buffalo, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Dose Level 1: Dose Level 1 Entinostat (3 mg, every 2 weeks, PO) Aldesleukin (600,000 IU/kg, every 8hrs, IV)
- Phase I Dose Level 2; Phase 2 Dose Level 2: Dose Level 2 Entinostat (5 mg, every 2 weeks, PO) Aldesleukin (600,000 IU/kg, every 8hrs, IV)
Period: Overall Study
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level 2 | Phase 2 Dose Level 2
Started | 3 | 8 | 36
Completed | 3 | 6 | 33
Not Completed | 0 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Groups:
- Dose Level 1: Dose Level 1 Entinostat (3 mg, every 2 weeks, PO) Aldesleukin (600,000 IU/kg, every 8hrs, IV)
- Dose Level 2: Dose Level 2 Entinostat (5 mg, every 2 weeks, PO) Aldesleukin (600,000 IU/kg, every 8hrs, IV)
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Total
Number analyzed (Participants) | 3 | 44 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (14.73) | 55.64 (8.35) | 55.53 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 7 | 7
  Male | 3 | 37 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 39 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicities of Entinostat When Combined With Aldesleukin Within the Phase I
Description: Number of dose-limiting toxicities of entinostat when combined with aldesleukin within the Phase I MEASUREMENT OF EFFECT Patients underwent CT scans at week 11 (+/- 7 days) of each cycle during aldesleukin administration and then every 8-12 weeks (+/- 2 weeks). Response Evaluation Criteria in Solid Tumors (RECIST V.1.0)
Time Frame: 84 days
Population: All treated and eligible Phase 1 patients
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 3 | 8
Participants | 0 | 0

2. Primary Outcome: Overall Response Rate (Complete Plus Partial) (Phase II)
Description: The proportion of patients who have a partial or complete response to treatment evaluated by RECIST V.1.0 criteria.
  MEASUREMENT OF EFFECT Patients underwent CT scans at week 11 (+/- 7 days) of each cycle during aldesleukin administration and then every 8-12 weeks (+/- 2 weeks). Response Evaluation Criteria in Solid Tumors (RECIST V.1.0)
Time Frame: Up to 12 months
Population: All Phase II treated and eligible patients
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- Treatment (Entinostat, Aldesleukin): Patients receive entinostat PO every 2 weeks beginning on day -14 and high-dose aldesleukin IV every 8 hours on days 1-5 and 15-19. Cycles repeat every 84 days* in the absence of disease progression or unacceptable toxicity.
  NOTE: *Patients with evidence of tumor shrinkage may receive up to 3 cycles of high-dose aldesleukin therapy. Patients with stable disease by RECIST version 1.0 criteria, but without evidence of tumor shrinkage after two cycles will receive only entinostat until disease progression is documented.
  Aldesleukin: Given IV
  Computed Tomography: Undergo FDG-PET/CT
  Entinostat: Given PO
  Fludeoxyglucose F-18: Undergo FDG-PET/CT
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Positron Emission Tomography: Undergo FDG-PET/CT
Arm/Group | Treatment (Entinostat, Aldesleukin)
Number analyzed (Participants) | 36
Proportion of participants | .39 [.26 to .54]

3. Secondary Outcome: Incidence of Toxicity (Phase I)
Description: Count of participants with grade 4 toxicity. The frequency and grade of toxicities will be tabulated for each dose level.
Time Frame: 84 days
Population: All Phase I patients
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 3 | 8
Participants | 1 | 0

4. Secondary Outcome: Progression-free Survival
Description: The median progression-free survival (PFS) was estimated using standard Kaplan-Meier methods, where estimates of the median were obtained with 95% confidence intervals (CIs). PFS was defined as the time from the start of treatment to progression or death due to any cause or last follow-up, patients who did not progress or die were censored.
  MEASUREMENT OF EFFECT Patients underwent CT scans at week 11 (+/- 7 days) of each cycle during aldesleukin administration and then every 8-12 weeks (+/- 2 weeks). Response Evaluation Criteria in Solid Tumors (RECIST V.1.0)
Time Frame: up to 12-months after the last subject enrolls
Population: All Phase 2 patients. PFS only assessed for Phase 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Entinostat, Aldesleukin)
Number analyzed (Participants) | 36
months | 14.0 [6 to NA] — Upper limit not reached

5. Secondary Outcome: Overall Survival
Description: The 3-year overall survival (OS) rate was estimated using standard Kaplan-Meier methods, where estimates of the median were obtained with 95% confidence intervals (CIs). OS was defined as the time from the start of treatment to death due to any cause or last follow-up, patients who did not die were censored.
Time Frame: up to 12-months after the last subject enrolls
Population: All Phase 2 patients. Overall Survival only assessed for Phase 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Entinostat, Aldesleukin)
Number analyzed (Participants) | 36
percentage of participants | 82.1 [62 to 93]

6. Secondary Outcome: Time-to-tumor Progression
Description: The median time to tumor progression (TTP) was estimated using standard Kaplan-Meier methods, where estimates of the median were obtained with 95% confidence intervals (CIs). TTP was defined as the time from the start of treatment to progression or last follow-up. Patients that did not progress were censored.
Time Frame: up to 12-months after the last subject enrolls
Population: All Phase 2 patients.TTP only assessed for Phase 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Entinostat, Aldesleukin)
Number analyzed (Participants) | 36
months | 14 [6.0 to NA] — Upper limit not reached

7. Secondary Outcome: Incidence of Toxicities
Description: The number of participants with serious adverse events.
Time Frame: Up to 30 days
Population: All Phase 2 patients. Toxicities only assessed for Phase 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Entinostat, Aldesleukin)
Number analyzed (Participants) | 36
Participants | 9

8. Secondary Outcome: Changes in the Level of Specific T Lymphocytes
Description: Mean percent change from baseline of T lymphocytes.
Time Frame: Baseline to approximately 4 weeks post-treatment, up to 1 year
Population: All treated and evaluable patients
Measure: Mean (Standard Deviation); unit: percentage of cells count
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 1 | 35
percentage of cells count | 26.3 (NA) — only 1 obsevation | 10.5 (70.8)

9. Secondary Outcome: Changes in Tumor Metabolisms by FDG Positron Emission Tomography (PET)/Computed Tomography (CT) Scan
Description: For binary predictors, the sensitivity and specificity with 95% confidence intervals will be reported. T tests will be used to compare the mean change between responders and non-responders. If there are sufficient numbers of responders, partial responders and non-responders an ANOVA will be used to compare changes in these three groups. If complete data are obtained for CD4+CD25^hi T cells at multiple time points post treatment, repeated measures ANOVA will be performed to evaluate data for trends over time.
Time Frame: Baseline to approximately 5 weeks post-treatment
Population: Data for this outcome was not collected. The investigator transferred from Hopkins to Roswell Park and the data for this outcome was not collected.
Arm/Group | Treatment (Entinostat, Aldesleukin)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the start date of intervention until 30 days after the last intervention, up to 1 year
Arm/Group | Dose Level 1 | Dose Level 2
All-Cause Mortality (participants affected / at risk) | 3/3 | 6/44
Serious Adverse Events (participants affected / at risk) | 0/3 | 9/44
Other Adverse Events (participants affected / at risk) | 1/3 | 35/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=44)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
White blood cell count (Investigations) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=44)
Anaemia (Blood and lymphatic system disorders) | 1 (3) | 27 (117)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 6 (9)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (3)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 3 (3)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 12 (18)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 9 (22)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 3 (3)
Dry eye (Eye disorders) | 0 (0) | 3 (4)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (5)
Constipation (Gastrointestinal disorders) | 0 (0) | 14 (24)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 9 (13)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 5 (6)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (2)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 30 (83)
Oral pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 23 (43)
Chest discomfort (General disorders) | 0 (0) | 3 (4)
Chest pain (General disorders) | 0 (0) | 2 (2)
Chills (General disorders) | 1 (1) | 21 (51)
Fatigue (General disorders) | 1 (5) | 32 (97)
Generalised oedema (General disorders) | 0 (0) | 1 (2)
Influenza like illness (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 2 (3)
Mucosal inflammation (General disorders) | 1 (1) | 2 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 8 (15)
Oedema peripheral (General disorders) | 1 (1) | 9 (17)
Pain (General disorders) | 0 (0) | 1 (1)
Polyp (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (4) | 23 (83)
Xerosis (General disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 6 (12)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Scrotal infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (2)
Tooth infection (Infections and infestations) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (2)
Adjusted calcium (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase decreased (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 6 (7)
Aspartate aminotransferase (Investigations) | 0 (0) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3)
Blood albumin (Investigations) | 0 (0) | 1 (2)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (5)
Blood bilirubin (Investigations) | 1 (4) | 20 (62)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine (Investigations) | 1 (3) | 2 (4)
Blood lactate dehydrogenase decreased (Investigations) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Haemoglobin (Investigations) | 1 (3) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (2) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 6 (7)
Lymphocyte count (Investigations) | 1 (1) | 18 (82)
Neutrophil count (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 8 (21)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 9 (25)
White blood cell count (Investigations) | 1 (5) | 19 (58)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 23 (46)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 25 (61)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (3) | 11 (15)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 7 (20)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 7 (8)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (5) | 28 (126)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (8) | 27 (154)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 11 (18)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 12 (34)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (4) | 23 (73)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (3) | 27 (123)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (8)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 11 (15)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 5 (6)
Dysgeusia (Nervous system disorders) | 0 (0) | 10 (16)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 13 (32)
Lethargy (Nervous system disorders) | 0 (0) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 3 (4)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (3)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 6 (8)
Confusional state (Psychiatric disorders) | 0 (0) | 15 (23)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 9 (14)
Hallucination (Psychiatric disorders) | 0 (0) | 2 (4)
Insomnia (Psychiatric disorders) | 1 (1) | 7 (12)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 6 (15)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 2 (2)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 6 (8)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 5 (7)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 12 (21)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 23 (53)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (10)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 13 (20)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 21 (32)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
Central venous catheterisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 4 (5)
Flushing (Vascular disorders) | 1 (3) | 10 (22)
Hypertension (Vascular disorders) | 1 (1) | 5 (7)
Hypotension (Vascular disorders) | 1 (3) | 26 (73)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/78/NCT01038778/Prot_SAP_000.pdf